CLINICAL TRIAL: NCT00687102
Title: Effects of Selective Estrogen Receptor Modulators on Cognitive Aging: Cognition in the Study of Tamoxifen and Raloxifene
Brief Title: Cognition in the Study of Tamoxifen and Raloxifene
Acronym: Co-STAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wake Forest University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IA0132; 1R13AG020218-01 (NIH); NCT00571857 (obsolete NCT alias)
Record Dates: First submitted 2008-05-28; First posted 2008-05-30 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Cognition; Aging
Keywords: breast cancer; Tamoxifen; Raloxifene; hormone therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Raloxifene Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Star participants assigned to Tamoxifen (Experimental): Participants in the parent study, STAR assigned to Tamoxifen who were 65 or older at time of enrollment.
  Interventions: Drug: tamoxifen
- Star participants assigned to Raloxifene (Experimental): Participants in the parent study, STAR assigned to Raloxifene who were 65 or older at time of enrollment.
  Interventions: Drug: raloxifene

INTERVENTIONS:
Drug: tamoxifen — oral tamoxifen plus placebo daily for 5 years
  Other Names: Nolvadex
  Arms: Star participants assigned to Tamoxifen
Drug: raloxifene — oral raloxifene plus placebo daily for 5 years
  Other Names: Evista, Keoxifene
  Arms: Star participants assigned to Raloxifene

SUMMARY:
The purpose of this study is to assess the effects of tamoxifen and raloxifene on cognitive aging in selected cognitively-healthy women.

DETAILED DESCRIPTION:
Recent reports indicate that hormone therapy (HT) may have a protective effect on the aging brain. Although previous studies have examined the effects of HT on age-related cognitive changes, there is little information on the effect of a new class of estrogenic agents, selective estrogen receptor modulators (SERMs), on cognitive aging. The two most commonly prescribed SERMs are tamoxifen, for treatment and prevention of breast cancer, and raloxifene, for maintaining bone density. In the face of potential widespread use of SERMs in healthy women, information on the effects of these agents on memory and other cognitive functions is essential.

The principal goals of Co-STAR are to compare the effects of tamoxifen and raloxifene

* on age-associated declines in measures of verbal and nonverbal memory in women over age 65
* other cognitive abilities and mood
* with those resulting from more common forms of HT, specifically ET (conjugated equine estrogen) and ET plus progesterone

Co-STAR results will be compared to results from the Women's Health Initiative Study of Cognitive Aging (WHISCA), a study involving 6-year longitudinal assessment of cognitive outcomes in 2969 women randomly assigned to receive active treatment (Premarin or Premarin plus medroxyprogesterone acetate) or placebo. A comparison of the Co-STAR treatment groups with the group of WHISCA participants receiving placebo will provide insights into the effects of SERMs relative to no treatment. A comparison of the Co-STAR treatment groups with WHISCA treatment groups receiving ET or ET plus progesterone will provide insights into the effects of SERMs relative to common HT treatments.

Co-STAR participants will be recruited from The National Cancer Institute's (NCI) Study of Tamoxifen and Raloxifene (STAR) NCT00003906, a multi-center, 5-year, randomized clinical trial among 22,000 women at increased risk for breast cancer, to compare the effects of tamoxifen and raloxifene on risk for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women enrolled in STAR trial at a site participating in Co-STAR
* 65 years of age or older
* Have been randomized into STAR but have not started taking the study drug OR enrolled in STAR for a minimum of one year
* Have not been diagnosed with dementia
* Have signed a separate consent document for the Co-STAR Study
* Previous diagnoses of chronic neurologic disease (Parkinson's disease, stroke, epilepsy, multiple sclerosis), history of head injury, depression, alcohol addiction, drug addiction, and other neurologic or psychiatric conditions will be recorded but will not serve as exclusion factors for this study

Exclusion Criteria:

* Not enrolled in the STAR Trial
* Younger than 65 years of age
* Diagnosed with dementia

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1498 (Actual)
Dates: Start 2001-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sally A. Shumaker, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (134):
- United States (127):
  - CCOP Western Regional, Phoenix, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - Naval Hospital Camp Pendleton, Camp Pendleton, California
  - City of Hope National Medical Center, Duarte, California
  - Hematology Oncology Consultants, Duarte, California
  - Southern Nevada Cancer Research Foundation, Duarte, California
  - Virginia K. Crosson Cancer Center, Fullerton, California
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - Valley Tumor Medical Group, Lancaster, California
  - Kaiser Permanente Division of Research, Oakland, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - North Valley Breast Clinic, Redding, California
  - Kaiser Permanente Oncology Research, San Diego, California
  - Naval Medical Center San Diego, San Diego, California
  - Cancer Foundation of Santa Barbara, Santa Barbara, California
  - Kaiser Permanente, Woodland Hills, Woodland Hills, California
  - Penrose Cancer Center, Colorado Springs, Colorado
  - Colorado Cancer Research Program, Denver, Colorado
  - St. Mary-Corwin Medical Center, Pueblo, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Lawrence & Memorial Hospital, New London, Connecticut
  - Christiana Care Health Services, Newark, Delaware
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - H. Lee Moffitt Cancer Center and Research Center, Tampa, Florida
  - Memorial Medical Center, Savannah, Georgia
  - University of Hawaii, Honolulu, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - SwedishAmerican Hospital Regional Cancer Ctr, Rockford, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Center for Cancer Care at Goshen Health Systems, Goshen, Indiana
  - Community Hospital, Munster, Indiana
  - CCOP,Northern Indiana Research Consortium, South Bend, Indiana
  - Genesis Medical Center, Davenport, Iowa
  - Finely Hospital, Wendt Regional Cancer Center, Dubuque, Iowa
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - The Harry and Jeanette Weinberg Cancer Institute at Franklin Square, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Berkshire Hematology Oncology, P.C., Pittsfield, Massachusetts
  - Genesys Hurley Cancer Institute, Ann Arbor, Michigan
  - Genesys Regional Medical Center, Ann Arbor, Michigan
  - Oakwood Healthcare System, Ann Arbor, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - St. John Hospital and Medical Center, Ann Arbor, Michigan
  - Battle Creek Health Systems, Battle Creek, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - McLaren Regional Medical Center, Flint, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Kalamazoo, Kalamazoo, Michigan
  - Michigan State University, Lansing, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - Mercy Memorial Hospital Cancer Center, Monroe, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Luke's Hospital, Duluth, Minnesota
  - Duluth Clinic, Duluth, Minnesota
  - Hennepin Consortium, Minneapolis, Minnesota
  - Metro-Minnesota, Saint Louis Park, Minnesota
  - Hematology & Oncology Associates Ltd, Tupelo, Mississippi
  - Ellis Fischel Cancer Center, Columbia, Missouri
  - St John's Regional Medical Center Cancer Center, Joplin, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - St John's Health System, Springfield, Missouri
  - Alvin J Siteman Cancer Center at Barnes-Jewish Hosp & Washington U Sch of Med, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Montana Cancer Consortium, Billings, Montana
  - Great Falls Clinic, LLP, Great Falls, Montana
  - Good Samaritan Health Systems, Kearney, Nebraska
  - Cancer Resource Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Cancer Center, Omaha, Omaha, Nebraska
  - Riverview Medical Center, Red Bank, New Jersey
  - Roswell Park/Western New York STAR Consortium, Buffalo, New York
  - Bassett Healthcare, Cooperstown, New York
  - Hematology-Oncology Associates of CNY, East Syracuse, New York
  - Vassar Brothers Hospital, Poughkeepsie, New York
  - University of Rochester Cancer Center, Rochester, New York
  - University Healthcare System, Syracuse, New York
  - Presbyterian Hospital, Charlotte, North Carolina
  - Blumenthal Cancer Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cape Fear Valley Medical Center, Fayetteville, North Carolina
  - Gaston Memorial Hospital, Gastonia, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Forsyth Regional Cancer Center, Winston-Salem, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Kaiser Permanente Ohio, Bedford, Ohio
  - Ireland Cancer Center at Case Western Reserve University, Cleveland, Ohio
  - CCOP Columbus, Columbus, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Fulton County Health Center, Toledo, Ohio
  - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Columbia River Oncology Program, Portland, Oregon
  - Kaiser Permanente Center for Health Research (Oncology Research), Portland, Oregon
  - UPMC/UPCI/Magee Women's Hospital, Pittsburgh, Pennsylvania
  - Mercy Cancer Center, Scranton, Scranton, Pennsylvania
  - York Cancer Center, York, Pennsylvania
  - Roper Hospital, Charleston, South Carolina
  - Palmetto Richland Memorial Hospital, Columbia, South Carolina
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Sioux Valley Clinic Oncology, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Methodist Hospitals of Dallas, Dallas, Texas
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - Baylor-Sammons Cancer Center, Dallas, Texas
  - UT Southwestern Center for Breast Care, Dallas, Texas
  - Baylor Medical Center at Garland, Garland, Texas
  - Breast Care Center at Baylor College of Medicine/Methodist Hospital, Houston, Texas
  - University of Texas M. D. Anderson Cancer Center, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Southwest Cancer Center, Lubbock, Texas
  - Baylor Regional Medical Center, Plano, Texas
  - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah
  - Danville Hematology & Oncology, Inc., Danville, Virginia
  - Olympic Hematology and Oncology Associates, Bremerton, Washington
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge Cancer Center, Yakima, Washington
  - Marshfield Clinic, Marshfield, Wisconsin
- Canada (7):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - UBC-Vancouver Hospital & Health Science Center, Vancouver, British Columbia
  - CancerCare Manitoba, Winnepeg, Manitoba
  - Women's Breast Health Centre, Ottawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Regional Cancer Care Clinical Trials, Thunder Bay, Ontario
  - North York General Hospital, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maki PM, Zonderman AB, Resnick SM. Enhanced verbal memory in nondemented elderly women receiving hormone-replacement therapy. Am J Psychiatry. 2001 Feb;158(2):227-33. doi: 10.1176/appi.ajp.158.2.227. PMID 11156805
- [Background] Resnick SM, Metter EJ, Zonderman AB. Estrogen replacement therapy and longitudinal decline in visual memory. A possible protective effect? Neurology. 1997 Dec;49(6):1491-7. doi: 10.1212/wnl.49.6.1491. PMID 9409335
- [Background] Resnick SM, Maki PM, Golski S, Kraut MA, Zonderman AB. Effects of estrogen replacement therapy on PET cerebral blood flow and neuropsychological performance. Horm Behav. 1998 Oct;34(2):171-82. doi: 10.1006/hbeh.1998.1476. PMID 9799627

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Co-STAR enrolled 1,498 women assigned in the STAR trial aged 65 years and older and no diagnosis of dementia. All participants were fluent in English and provided written informed consent for the Co-STAR study. Enrollment began in October 2001, 18 months after STAR enrollment started and continued until the unmasking of STAR in June 2006.
Period: Overall Study
Arm/Group | Star Participants Assigned to Tamoxifen | Star Participants Assigned to Raloxifene
Started | 733 | 765
Completed | 733 | 765
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Star Participants Assigned to Tamoxifen | Star Participants Assigned to Raloxifene | Total
Number analyzed (Participants) | 733 | 765 | 1498
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 733 | 765 | 1498
Sex: Female, Male [Count of Participants; unit: Participants] — This study was designed to recruit female participants only.
  Participants
    Female | 733 | 765 | 1498
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 685 | 715 | 1400
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 48 | 50 | 98

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline on the the Benton Visual Retention Test Scores by Treatment Group
Description: Mean Change From Baseline on the Benton Visual Retention (BVRT) Test scores. Adjusted for age, ethnicity, education, and baseline measure, for participants with true baseline measures.
  The BVRT measures short term visual memory and visuo-constructional abilities. Each of 10 designs was presented one at a time for 10 seconds, and immediately after the design was withdrawn, the participant was instructed to draw it from memory on a blank sheet of paper. The score on the BVRT is the total number of errors, 0-26 represents the total number of theoretically possible errors. Lower score denotes better outcomes.
Time Frame: Baseline and 3 Years
Population: Women who were randomly assigned in STAR were age 65 years and older, were not diagnosed with dementia, and were enrolled onto the Cognition in the Study of Tamoxifen and Raloxifene (Co-STAR) trial.
Measure: Mean (Standard Error); unit: Number of errors
Arm/Group | Star Participants Assigned to Tamoxifen | Star Participants Assigned to Raloxifene
Number analyzed (Participants) | 83 | 93
Number of errors | -0.73 (0.34) | -1.41 (0.32)

2. Primary Outcome: Mean Change From Baseline on the the California Verbal Learning Test Scores by Treatment Group
Description: Adjusted for age, ethnicity, education, and baseline measure, for participants with true baseline measures.
  The experimenter reads a list of 16 nouns aloud, at one-second intervals, in fixed order, over 3 learning trials (list A) . After each trial, the subject is asked to recall as many words as they can in any order (i.e., free recall) given a score 0-16 each. Total range as the sum of the 3 learning trials: 0 - 48. Participants were asked to recall a second interference list (List B) with a score range of 0-16. Free recall of list A are tested immediately after list B (short-delay) Total range 0- 16 , and again after 20 minutes (long-delay) 0-16. Each part of the scale is reported separately as Total List A trials, Total List B trials, Short-delay free recall, and Long-delay free recall.
Time Frame: Baseline and 3 Years
Population: as for outcome 1
Measure: Mean (Standard Error); unit: correct responses
Arm/Group | Star Participants Assigned to Tamoxifen | Star Participants Assigned to Raloxifene
Number analyzed (Participants) | 83 | 93
correct responses
  Total List A trials | -3.31 (0.50) | -1.89 (0.48)
  Total List B trials | -1.56 (0.19) | -1.74 (0.18)
  Short-delay free recall | -0.96 (0.25) | -0.36 (0.24)
  Long-delay free recall | -0.23 (0.25) | 0.10 (0.24)

3. Secondary Outcome: Mean Change From Baseline on the Letter Fluency and Semantic Fluency Scores by Treatment Group
Description: Mean Change From Baseline on the Letter Fluency Test scores. Adjusted for age, ethnicity, education, and baseline measure, for participants with true baseline measures.
  Measures cognitive function. In this test, the participant names as many words as possible in 1 minute, beginning with each letter for letter fluency (F, A, and S) and category for semantic fluency (fruits and vegetables). To score the administrator, counts up the total number letters or words that the individual is able to produce. The score minimum would be 0 and the maximum would be the total of correct items named within 1 minute. Higher scores represent better outcomes.
Time Frame: Baseline and 3 Years
Population: as for outcome 1
Measure: Mean (Standard Error); unit: change in number of words
Arm/Group | Star Participants Assigned to Tamoxifen | Star Participants Assigned to Raloxifene
Number analyzed (Participants) | 83 | 93
change in number of words
  Letter Fluency | 1.29 (0.75) | 1.51 (0.71)
  Semantic Fluency | -.51 (.50) | -.56 (.47)

4. Secondary Outcome: Mean Change From Baseline on Digit Span Test Scores by Treatment Group
Description: Mean Change From Baseline on the Digit Span Test - Digits Forward and Digits backward Test scores. Adjusted for age, ethnicity, education, and baseline measure, for participants with true baseline measures.
  Measures reasoning, verbal ability, and memory. The participant is asked to provide immediate recall of a series of digits in forward and backward sequences. The individual's score is the total number of items correctly repeated forwards or backwards. Total range 0 - 14, higher results denotes a better outcome.
Time Frame: Baseline and 3 Years
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Star Participants Assigned to Tamoxifen | Star Participants Assigned to Raloxifene
Number analyzed (Participants) | 83 | 93
units on a scale
  Digits Forward | -0.02 (0.18) | -0.08 (0.17)
  Digits Backward | -0.16 (0.17) | -0.27 (0.16)

5. Secondary Outcome: Mean Change From Baseline on Card Rotations Test Scores by Treatment Group
Description: Mean Change From Baseline on the Card Rotations Test scores. Adjusted for age, ethnicity, education, and baseline measure, for participants with true baseline measures.
  Measures the ability to mentally manipulate figures in two and three-dimensions. On each of 28 trials, participants view sample line drawings of a geometric figure and 8 alterations representing 2 or 3-dimensional rotations of the drawing. Participants are asked to identify alternatives that show the sample in 2-D but not in 3-D. Total range 0 - 160 and the number of incorrect/correct responses is measure. Higher number of correct answers is a better outcome.
Time Frame: Baseline and 3 Years
Population: as for outcome 1
Measure: Mean (Standard Error); unit: correct responses
Arm/Group | Star Participants Assigned to Tamoxifen | Star Participants Assigned to Raloxifene
Number analyzed (Participants) | 83 | 93
correct responses | 6.10 (1.97) | 5.40 (1.86)

6. Secondary Outcome: Mean Change From Baseline on the Finger Tapping Test Scores by Treatment Group
Description: Mean Change From Baseline on the the Finger Tapping Test scores. Adjusted for age, ethnicity, education, and baseline measure, for participants with true baseline measures.
  Measures motor speed, coordination, attention, alertness, slowing of responses, and motor control. In this test of motor speed and dexterity participants are asked to depress a lever as many times as possible in each of 7, 10-second trials, first with the right hand and next with the left hand. The highest and lowest scores are dropped; the score is the average of the remaining five trials for each hand.Higher scores represent better outcomes.
Time Frame: Baseline and 3 Years
Population: as for outcome 1
Measure: Mean (Standard Error); unit: finger taps
Arm/Group | Star Participants Assigned to Tamoxifen | Star Participants Assigned to Raloxifene
Number analyzed (Participants) | 83 | 93
finger taps
  Fine Tapping, Dominant | 0.26 (0.65) | -0.04 (0.63)
  Fine Tapping, Non-Dominant | -0.18 (0.50) | -0.45 (0.48)

7. Secondary Outcome: Mean Change From Baseline on the Positive and Negative Affect Schedule Scores by Treatment Group
Description: Mean Change From Baseline on the Positive and Negative Affect Schedule (PANAS). Adjusted for age, ethnicity, education, and baseline measure, for participants with true baseline measures.
  Measures positive and negative affect. Mood is assessed with the PANAS, a list of ten pleasant mood states (e.g., interested, proud, inspired) and ten unpleasant mood states (e.g., irritable, guilty, jittery). Respondents are asked to rate on a 5-point scale (1 being "very slightly or not at all" and 5 being "extremely") the extent to which they have experienced each mood during a specific time frame. Ratings for each item can range from 0 to 4 with total scores for positive affect and negative affect subscales ranging from 0 to 40. For positive affect, higher scores denote higher levels of positive affect and for negative affect, lower scores denote lower levels of negative affect.
Time Frame: Baseline and 3 Years
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Star Participants Assigned to Tamoxifen | Star Participants Assigned to Raloxifene
Number analyzed (Participants) | 83 | 93
units on a scale
  PANAS-positive | -0.10 (0.06) | -0.04 (0.05)
  PANAS-negative | 0.00 (0.06) | -0.06 (0.05)

8. Secondary Outcome: Mean Change From Baseline on the Geriatric Depression Scale Scores by Treatment Group
Description: Mean Change From Baseline on the Geriatric Depression Scale. Adjusted for age, ethnicity, education, and baseline measure, for participants with true baseline measures.
  Measures depression in older adults. Mood is also assessed with the 15-item short form of the GDS which measures non-somatic features of depressed mood. Participants indicate the presence or absence of each symptom. The GDS-SF score is the total number of positive depressive items. Score range is 0-15, with 0-4 denoting better outcomes and a score of 5 and above denoting worse outcomes (depression).
Time Frame: Baseline and 3 Years
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Star Participants Assigned to Tamoxifen | Star Participants Assigned to Raloxifene
Number analyzed (Participants) | 83 | 93
units on a scale | 0.57 (0.19) | 0.13 (0.18)

ADVERSE EVENTS:
Time Frame: 4 years, 8 months
Arm/Group | Star Participants Assigned to Tamoxifen | Star Participants Assigned to Raloxifene
Serious Adverse Events (participants affected / at risk) | 0/733 | 0/765
Other Adverse Events (participants affected / at risk) | 0/733 | 0/765

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No